CLINICAL TRIAL: NCT04161807
Title: Efficacy and Safety of Nerivio™, a Remote Electrical Neuromodulation Device, for Acute Treatment of Migraine in People With Chronic Migraine: an Open Label, Single Arm, Multicenter Study
Brief Title: Efficacy and Safety of Nerivio™ for Acute Treatment of Migraine in People With Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCH005
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2019-12

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Nerivio device treatment (Experimental): participant will receive the Nerivio device for treating their migraine attacks. Treatment will be perform as soon as the participant feel that the migraine attack started
  Interventions: Device: Nerivio

INTERVENTIONS:
Device: Nerivio — The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application.

SUMMARY:
This study is intended to evaluate the efficacy and safety of Nerivio, an FDA-authorized remote electrical neuromodulation (REN) device for the acute treatment of migraine, for the acute treatment of migraine in people with chronic migraine. The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The study duration consists of a 4 weeks of active treatment with the device in about 40 patients.

DETAILED DESCRIPTION:
This open label study includes up to 2 visits. The enrollment and device training may occur in 2 separate visits.

First visit - The first visit will include screening, enrollment and training on the application and device.

Treatment phase - Participants will be instructed to use the device for the treatment of qualifying migraine headaches (see below) as soon as possible and always within 60 minutes of onset during a period of up to 4 weeks. Participants will be instructed to use the device with the intensity level identified during the device training visit (and adjust as necessary) and make sure the stimulation is perceptible but not painful. Participants will be instructed to avoid taking rescue medications within 2 hours post-treatment. If medications are used, participants will be instructed to record in the app when and which medication was taken at 2- and 24-hours post treatment. The participants will use the app to record pain intensity levels, the presence/absence of aura and associated migraine symptoms (nausea, photophobia, phonophobia, and allodynia l) as well as rate their stress level and functional disability at baseline, 2- and 24-hours post-treatment. At the beginning of each treatment, participants will also be asked to report the time elapsed from attack onset. Adverse events will be reported throughout this phase of the study directly to the site staff.

Participants who do not achieve satisfactory relief at 2 hours post-treatment may treat again with the Nerivio™ device or may treat with usual care at that time or any time thereafter if the headache does not resolve. Participants will also be able to treat headache recurrence with the device. Migraine headaches that are not treated with the device may be treated with usual care.

The first reported treatment will be considered a "training" treatment, aimed to verify that the participants use the device properly, and will only be included in the safety analysis. The efficacy evaluation will be performed on the first treatment of a qualifying attack (see below) following the training treatment (hereby termed "test treatment").

Second (final) visit - End of study:

Participants will return to the clinic following the end of the treatment phase, at which time they will return the device. The participants will have the option of returning the device by mail instead of an on-site visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18-75 years old.
2. Participants meeting the ICHD-3 diagnostic criteria for chronic migraine
3. Participants have personal access to a smartphone
4. Participants must be able and willing to comply with the protocol
5. Participants must be able and willing to provide written informed consent

Exclusion Criteria:

1. Participants with an implanted electrical and/or neurostimulator device (e.g. cardiac pacemaker, cochlear implant).
2. Participants with congestive heart failure (CHF), severe cardiac or cerebrovascular disease.
3. Participants with uncontrolled epilepsy.
4. Lack of efficacy, after an adequate therapeutic trial, of at least two migraine specific acute medications
5. Change in migraine preventive medications (type or dose) in the last two months prior to recruitment and/or during the study
6. Pregnant, trying to get pregnant or breastfeeding female participants
7. Subjects participating in any other interventional clinical study.
8. Participants without basic cognitive and motor skills needed to operate a smartphone
9. Participants with other significant pain, medical or psychological problems that in the opinion of the investigator may confound the study assessments
10. Participants who have previous experience with the device

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wright, Principal Investigator — Nuvance Health
Locations (2):
- Health Quest Medical Practice, PC, Lagrangeville, New York, United States
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nierenburg H, Vieira JR, Lev N, Lin T, Harris D, Vizel M, Ironi A, Lewis B, Wright P. Remote Electrical Neuromodulation for the Acute Treatment of Migraine in Patients with Chronic Migraine: An Open-Label Pilot Study. Pain Ther. 2020 Dec;9(2):531-543. doi: 10.1007/s40122-020-00185-1. Epub 2020 Jul 9. PMID 32648205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from September 18, 2019 to February 18, 2020. . Study sites were Nuvance health (Poughkeepsie, NY) and Meir Medical center (Kefar Sava, Israel). 42 patients were enrolled and received a device. Two participants withdrew from the study.
  All participants completed at least one treatment (the training treatment) and 38 participants completed the test treatment, forming the final analysis set.
Period: Overall Study
Arm/Group | Nerivio Device Treatment
Started | 42
Completed | 38
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Performed only 1 treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
  Israel | 12
Average number of headache days per month [Mean (Standard Deviation); unit: Days per month] | 21.5 (6.3)
Average number of migraine headache das per month [Mean (Standard Deviation); unit: Days per month] | 18.3 (6.6)
Use of preventive medication [Count of Participants; unit: Participants] | 27

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Reduction of Migraine Headache at 2 Hours Post Treatment
Description: The proportion of participants reporting pain relief at 2 hours post-treatment without the use of rescue medication following the test treatment . Pain relief is defined as an improvement from severe or moderate pain to mild or no pain, or from mild pain to no pain.
Time Frame: 2 hours post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 38
Participants | 19

2. Secondary Outcome: Proportion of Participants With Pain Disappearance at 2 Hours Post Treatment
Description: The proportion of participants reporting freedom from migraine pain at 2 hours post-treatment without medications following the test treatment. Pain freedom is defined as an improvement from severe or moderate or mild pain to no pain
Time Frame: 2 hours post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 38
Participants | 10

3. Secondary Outcome: Proportion of Participants With Disappearance of Nausea and/or Vomiting at 2 Hours Post-treatment
Description: The proportion of participants reporting disappearance of nausea and/or vomiting at 2 hours post-treatment without rescue medications following the test treatment.
Time Frame: 2 hours post treatment
Population: only 17 participants reported nausea and/or vomiting at T=0 hours of the Test treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 17
Participants | 10

4. Secondary Outcome: Proportion of Participants With Disappearance of Photophobia at 2 Hours Post-treatment
Description: The proportion of participants reporting disappearance of photophobia at 2 hours post-treatment without rescue medications following the test treatment.
Time Frame: 2 hours post treatment
Population: only 24 participants reported photophobia at T=0 hours of the Test treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 24
Participants | 9

5. Secondary Outcome: Proportion of Participants With Disappearance of Phonophobia at 2 Hours Post-treatment
Description: The proportion of participants reporting disappearance phonophobia at 2 hours post-treatment without rescue medications following the test treatment.
Time Frame: 2 hours post treatment
Population: only 16 participants reported phonophobia at T=0 hours of the Test treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 16
Participants | 8

6. Other Pre Specified Outcome: Within-patient Consistency - Percentage of Participants With Reduction in Headache Pain in at Least 50% of Their Treatments
Description: Proportions of participants achieving pain relief at 2 hours in at least 50% of all their treatments (excluding the training treatment)
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 38
Participants | 27

7. Other Pre Specified Outcome: Within-patient Consistency - Percentage of Participants Free of Headache Pain in at Least 50% of Their Treatments
Description: Proportion of participants achieving pain free at 2 hours in at least 50% of all their treatments (excluding the training treatment)
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 38
Participants | 10

8. Other Pre Specified Outcome: Proportion of Participants With Improve Functional Disability at 2 Hours Post-treatment
Description: The proportion of participants achieving improvement of at least one grade in functional disability in the test treatment at 2 hours post-treatment with no use of rescue medication. the scale used was: (0) No limitation, (1) Some limitation, (2) Moderate limitation and (3) Severe limitation.
Time Frame: 2 hours post treatment
Population: Only 30 participants reported their function disability level at T=0 hours and T=2 hours for their test treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 30
Participants | 14

9. Other Pre Specified Outcome: Proportion of Participants With Improve Functional Disability at 24 Hours Post-treatment
Description: The proportion of participants achieving improvement of at least one grade in functional disability in the test treatment at 24 hours post-treatment with no use of rescue medication. the scale used was: (0) No limitation, (1) Some limitation, (2) Moderate limitation and (3) Severe limitation.
Time Frame: 24 hours post treatment
Population: Only 19 participants reported their function disability level at T=0 hours and T=24 hours for their test treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 19
Participants | 15

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Description: The Nerivio device is a neurostimulator and it is externally applied over the body.The Nerivio is accepted as a non-significant risk (NSR) device. In addition, as theexclusion criteria for the study leave out participant with electrical implant,congenital heart failure or epilepsy, the number of high risk participants is zero.
Arm/Group | Nerivio Device Treatment
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 1/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nerivio Device Treatment (N=42)
Tingling (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No limitations or caveats were reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT04161807/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT04161807/ICF_001.pdf